CLINICAL TRIAL: NCT02358694
Title: Safety and Tolerability of Serum-Derived Bovine Immunoglobulin in Children With Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: Safety and Tolerability of Serum Derived Bovine Immunoglobulin in Children With Diarrhea Predominant IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Hyams, MD, Chair, Pediatrics Gastroenterology, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBI-IBS-D
Record Dates: First submitted 2014-11-07; First posted 2015-02-09 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome
Keywords: IBS; IBS-D; SBI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Group (Experimental): Patients who weigh less than 40 Kg will receive 5 g daily (2.5 g PO BID) of Serum-derived bovine immunoglobulin/ protein isolate Patients who weigh 40 Kg or more will receive 10 g daily (5 g PO BID) of Serum-derived bovine immunoglobulin/ protein isolate
  Interventions: Dietary Supplement: Serum-Derived Bovine Immunoglobulin
- Placebo Arm (Placebo Comparator): The placebo group will receive a hydrolyzed gelatin protein for next 4 weeks on a daily basis.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Serum-Derived Bovine Immunoglobulin — Patients who weigh less than 40 Kg will receive Serum Derived Bovine Immunoglobulin -5 g daily (2.5 g PO BID) and patients who weigh 40 Kg or more will receive Serum Derived Bovine Immunoglobulin- 10 g daily (5 g PO BID)
  Other Names: SBI; Entera
  Arms: Active Treatment Group
Other: Placebo — Matching placebo packets will be supplied and will appear identical to SBI with respect to volume, appearance and taste.
  Patients who weigh less than 40 Kg will take one-half packet BID (2.5 g BID) Patients who weigh 40 Kg or more will take one packet BID (5 g PO BID).
  Arms: Placebo Arm

SUMMARY:
This study is being conducted to see if serum-derived bovine immunoglobulin/protein isolate (SBI) is safe and well tolerated in pediatric patients with IBS-D.

Main Hypothesis :Pediatric patients with IBS-D, who take SBI, will have no significant adverse events at 4 and 8 weeks and their quality of life will be better than the patients who receive placebo.

DETAILED DESCRIPTION:
The study will consist of four phases:

Screening Phase: screen the patients for 2 weeks prior to enrollment in the study to establish objective criteria of disease presence and severity. Patients will maintain a daily symptom dairy. At the end of screening phase, we will calculate their quality of life and symptom severity scores based on the information provided by the patients and their family. Patients with an average score of 1 or greater over 14 days for abdominal pain and stool consistency will be selected for the open label trial of SBI.

Open Label Treatment Phase: patients enrolled will receive 4 weeks of SBI along with QOL questionnaires to complete. If the patient's global assessment is that they have improved, or if review of their diaries shows an improvement in symptom severity scores (decrease in symptom severity score by > 30% from baseline), they will be eligible for the randomization phase.

Patients, who do not have any improvements during the first 4 weeks of SBI therapy, will not be randomized. If non-responders have worsening of symptoms, they will be prescribed rescue medications as per standard of care. If non-responders choose to continue to take SBI, they will be so allowed.

Randomization Phase: Patients who qualify for this phase will be randomized either to SBI or placebo. They will take their medication for 4 more weeks and complete their questionnaires, symptom as well as QOL. After this 4 week phase all patients will be offered the Open Label Extension Phase.

Open Label Extension Phase: All patients who enter this phase will be treated with SBI for another 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 8 years of age and < 18 years of age
* Patients with a diagnosis of IBS-D as per Rome III criteria
* Patients with normal laboratory work up (CBC, ESR, CRP, amylase, lipase, celiac panel, fecal occult blood)
* Patients with normal fecal calprotectin and lactose hydrogen breath test
* Patients off motility drugs, NSAIDs for at least 2 weeks prior to enrollment in the study
* Ability to complete the study
* Patients on stable doses or other medications for at least 4 weeks prior to enrollment

Exclusion Criteria:

* Patients with h/o other GI, hepatic, renal, cardiovascular, neurologic or hematological disorder
* Patients with family history of inflammatory bowel disease
* Patients with history of abdominal surgery
* Patient with history of drug or alcohol abuse
* Patient with a history of allergy to study related products (e.g. beef)
* Use of probiotics in the previous month
* Patients who used SBI in the past
* Patients with soy allergy/sensitivity

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Intervals from 0 to 4 weeks and from 4 to 8 weeks
  The ability of children to take SBI and related side effects

SECONDARY OUTCOMES:
Quality of Life Scores | Assessed at Day 0, 4 weeks and 8 weeks
  The proportion of subjects who achieve an improvement in their symptoms at the end of different study assessment times.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Rana, MD, Principal Investigator — Connecticut Childrens Medical Center
Locations (1):
- Connecticut Childrens Medical Center, Farmington, Connecticut, United States